CLINICAL TRIAL: NCT01518231
Title: Phase 1 Study of Autologous Peripheral Hematopoietic Stem Cell Transplantation in Ischemic Stroke
Brief Title: Autologous Hematopoietic Stem Cell Transplantation in Ischemic Stroke
Acronym: AHSCTIS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Hospital (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Yaguo Li, Yaguo Li, Zhejiang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhejiang Hospital
Record Dates: First submitted 2012-01-10; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Stroke
Keywords: stroke; hematopoietic stem cell transplantation
MeSH Terms: conditions — Stroke | interventions — Aspirin; Warfarin; Atorvastatin; Edaravone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cell transplantation (Experimental): The study group will not only be implanted with autologous hematopoietic stem cells, but also receive drug therapy.
  Interventions: Procedure: autologous hematopoiesis stem cell transplantation; Drug: Aspirin; Drug: Warfarin; Drug: Atorvastatin; Drug: Edaravone
- Convention therapy (No Intervention): The control group just receive drug therapy.
  Interventions: Drug: Aspirin; Drug: Warfarin; Drug: Atorvastatin; Drug: Edaravone

INTERVENTIONS:
Procedure: autologous hematopoiesis stem cell transplantation — Every participant will be transplanted with about 4 million autologous peripheral blood stem cell(CD34+) through cerebral artery.
  Arms: cell transplantation
Drug: Aspirin — aspirin 100mg,qd,po(patients with no fibrillation atrial)
  Arms: cell transplantation
Drug: Warfarin — warfarin 2~6mg,qd,po(patients with fibrillation atrial);
  Arms: cell transplantation
Drug: Atorvastatin — atorvastatin 20mg,qd,po
  Arms: cell transplantation
Drug: Edaravone — edaravone 30mg,bid,ivgtt.
  Arms: cell transplantation
Drug: Aspirin — aspirin 100mg,qd,po(patients with no fibrillation atrial)
  Arms: Convention therapy
Drug: Warfarin — warfarin 2~6mg,qd,po(patients with fibrillation atrial)
  Arms: Convention therapy
Drug: Atorvastatin — atorvastatin 20mg,qd,po
  Arms: Convention therapy
Drug: Edaravone — edaravone 30mg,bid,ivgtt
  Arms: Convention therapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of autologous peripheral hematopoietic stem cell transplantation in ischemic stroke.

DETAILED DESCRIPTION:
Stroke is among the main causes of mortality and disability of elderly population which still lack of efficient therapy. Stem sell transplantation provides a functional improvement after cerebral ischemia in rat models. Our study will recruit 40 ischemic stroke patients which will be divided into 2 groups (20 patients each): treatment group and control group. The former will be implanted with peripheral blood stem cell through anterior cerebral artery or middle cerebral artery (determined by the section of infarction) and receive convention stroke therapy. The latter only receive convention stroke therapy. The investigators expect that transplantation of the peripheral hematopoietic stem cell is safe and efficient to neurological recovery.

ELIGIBILITY:
Inclusion Criteria:

* aged 40~70
* no consciousness disorders
* internal carotid artery territory infarction
* stroke happened < 1 year
* with stable hemiplegia, but remain dependent in daily life
* SSS(Scandinavian Stroke Scale) < 40

Exclusion Criteria:

* pregnant women
* can't tolerate the test because of other disease, such as heart failure, liver failure, renal failure, abnormal blood coagulation, AIDS, combine other tumor or special condition

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in NIH-stroke scale (NIHSS) at 12 months | 1,3,6,12 months after cell transplantation

SECONDARY OUTCOMES:
Barthel index | 1,3,6,12 months after cell transplantation
perfusion magnetic resonance imaging scan | 1,3,6,12 months after cell transplantation
Modified Rankin Scale(mRS) | 3,6,12 months after cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Yaguo Li, master, Study Director — Zhejiang Hospital; Yumiao Zhou, master, Principal Investigator — Zhejiang Hospital
Locations (1):
- Yaguo Li, Hangzhou, Zhejiang, China